CLINICAL TRIAL: NCT02572778
Title: Establishment of Primary Patient-derived Xenograft Models of Tumor From Patients With Head and Neck Cancer for Preclinical Evaluation of Targeted Therapies.
Brief Title: Patient-derived Xenograft Models of Tumor From Patients With Head and Neck Cancer
Acronym: UCL-Xenog
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: UCL-ONCO2015-02
Record Dates: First submitted 2015-09-22; First posted 2015-10-09 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies of the tumor of the patients with squamous cell carcinoma of the head and neck
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Local biopsy in the tumor — A tumor biopsy of 0.5 cm2 or more will be collected from every patient during surgery or endoscopy after informed consent and if there is enough material after review by the pathologist.

SUMMARY:
The investigators want to have a collection of fresh primary or recurrent tumor tissue for establishment of patients-derived xenografts in order to:

generate a biobank of in vivo patient xenografts representing the different subgroups of tumors for head and neck cancer

* perform genetic and transcriptional profiling of the primary, metastatic tumors and xenograft tumors
* evaluate the efficacy of new targeted agents, whether or not in combination with standard treatment options
* evaluate biomarkers of drug sensitivity
* study primary and secondary (acquired) resistance in these models

ELIGIBILITY:
Inclusion Criteria:

* In the first phase, all patients with primary or recurrent/ metastatic disease of head and neck cancer can be included pre-operatively or before a tumor biopsy after obtaining informed consent
* Data on stage, grade, histology, adjuvant treatment, responses, relapse should be available
* Follow-up data should be available
* Patients with recurrent disease are allowed
* Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a primary advanced or recurrent head and neck tumor.
  * Inclusion preoperatively or before biopsy
  * Written informed consent prior to surgery or biopsy
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of the biomarkers of new cancer therapies for head and neck cancer on the patient-derived xenografts with immunohistochemistry (KI67) on FFPE (fixation followed by paraffin embedding) slides | 10 years
  Identification of the biomarkers of new cancer therapies for head and neck

SECONDARY OUTCOMES:
Characterization of the biomarkers of new cancer therapies for head and neck cancer on the patient-derived xenografts with genetic techniques | 10 years
  Characterization of the biomarkers of new cancer therapies for head and neck cancer on the patient-derived xenografts with genetic techniques

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Machiels, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium